CLINICAL TRIAL: NCT04414631
Title: Recombinant Human C1 Esterase Inhibitor (Conestat Alfa) in the Prevention of Severe SARS-CoV-2 Infection in Hospitalized Patients With COVID-19: a Randomized, Parallel-group, Open-label, Multi-center Pilot Trial (PROTECT-COVID-19).
Brief Title: Conestat Alfa in the Prevention of Severe SARS-CoV-2 Infection in Hospitalized Patients With COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Aim to enroll 120 patients deemed not sufficient to show a difference in the primary outcome measure. Standard of care treatment recently changed in Switzerland adding further heterogeneity to trial population when including future participants.
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Pharming Technologies B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-01252; me20Osthoff3
Record Dates: First submitted 2020-05-19; First posted 2020-06-04 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Coronavirus Infections
Keywords: Systemic hyperinflammation; cytokine storm; complement system; kinin-kallikrein system; C1 esterase inhibitor; Conestat alfa; Coronavirus Disease 19 (COVID-19); Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)
MeSH Terms: conditions — Coronavirus Infections; Cytokine Release Syndrome; Angioedemas, Hereditary; COVID-19 | interventions — conestat alfa

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, parallel-group, controlled, multi-center clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active treatment arm (Active Comparator): treatment with conestat alfa in addition to standarf of care
  Interventions: Drug: Conestat alfa
- Standard of care treatment arm (No Intervention): Standard of care treatment established at the centers

INTERVENTIONS:
Drug: Conestat alfa — Conestat alfa (8400 Units (U) followed by 4200 U every 8 hours, 9 administrations in total) will be administered as a slow intravenous injection (5-10 minutes) over a 72 hour period.
  Arms: active treatment arm

SUMMARY:
The aim of this study is to analyze if administration of conestat alfa for 72 hours in addition to standard of care (SOC) in patients hospitalized with non-critical SARS-CoV-2 pneumonia (WHO Ordinal Scale Score 3 or 4) reduces the risk of disease progression to Acute Lung Injury (ALI) and Acute Respiratory Distress Syndrome (ARDS).

DETAILED DESCRIPTION:
Systemic hyperinflammation is a hallmark of more severe stages of COVID-19 leading to acute respiratory distress syndrome, mechanical ventilation and ultimately death. In this stage, COVID-19 is associated with a decrease in suppressor and regulatory T cell counts and an extensive release of proinflammatory cytokines and biomarkers called a cytokine storm, which is thought to be the major driver of severe pneumonia caused by SARS-CoV-2. C1 esterase inhibitor (C1INH) is a member of the serpin superfamily of serine-protease inhibitors and is a strong inhibitor of the complement System (CS) and the kinin-kallikrein (KK) System. Conestat alfa is a recombinant human C1INH, that shares an identical protein structure with plasma-derived C1INH. The rationale of the current trial is based upon the following assumptions: In the context of COVID-19, conestat alfa treatment may 1) dampen uncontrolled complement activation and collateral lung damage and 2) reduce capillary leakage and subsequent pulmonary edema by direct inhibition of KK system. The aim of this study is to analyze administration of conestat alfa for 72 hours in addition to standard of care in patients hospitalized with non-critical SARS-CoV-2 pneumonia (WHO Ordinal Scale Score 3 or 4) and its association with clinical severity on day 7 after inclusion and the risk of disease progression to Acute Lung Injury (ALI) and Acute Respiratory Distress Syndrome (ARDS).

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* admitted to the hospital because of confirmed (by a positive SARS-CoV-2 PCR result) COVID-19 infection
* evidence of pulmonary involvement on CT scan or X-ray of the chest (e.g. ground glass opacities)
* symptom onset within the previous 10 days OR shortness of breath within the previous 5 days. Symptoms include fever or one respiratory symptom (patients presenting later may have already progressed to an inflammatory state that is potentially not amenable to C1INH treatment). Respiratory symptoms include cough, sore throat, hemoptysis, shortness of breath, runny nose, or chest pain.
* expected to remain an inpatient over the next three calender days from time of enrolment
* at least one additional risk factor for progression to mechanical ventilation: 1) arterial hypertension, 2) >50 years, 3) obesity (BMI>30.0 kg/m2), 4) cardiovascular disease, 5) chronic pulmonary disease, 7) chronic renal disease, 6) C-reactive protein of >35mg/L, 7) oxygen saturation at rest in ambient air of <94%. Cardiovascular disease includes a history of coronary artery disease, cerebrovascular disease, peripheral artery disease, rheumatic heart disease, congenital heart disease and of recent (< 3 months) deep vein thrombosis or pulmonary embolism. Chronic pulmonary disease includes a history of chronic obstructive pulmonary disease, asthma, occupational lung disease, interstitial lung disease or of pulmonary hypertension. Chronic renal disease is defined as a history of an estimated glomerular filtration rate (according to the Chronic Kidney Disease Epidemiology Collaboration equation) < 60ml/min/1.73 m2 for at least three months.

Exclusion Criteria:

* Contraindications to the class of drugs under study (C1 esterase inhibitor), e.g. known hypersensitivity or allergy to class of drugs or the investigational product
* Treatment with tocilizumab or another Il-6R or Il-6 inhibitor before enrolment
* History or suspicion of allergy to rabbits
* Women who are pregnant or breast feeding
* Active or planned treatment with any other complement inhibitor
* Liver cirrhosis (any Child-Pugh score)
* Incapacity or inability to provide informed consent
* Currently admitted to an ICU or expected admission within the next 24 hours
* Currently receiving invasive or non-invasive ventilation (with the exception of high-flow oxygen therapy).
* In the opinion of the treating time, death is deemed to be imminent and inevitable within the next 24 hours
* Participation in another study with investigational drug within the 30 days preceding and during the present study with the following exemptions: 1) participation in COVID-19 drug trials started at least 48 hours before admission (e.g. postexposure prophylaxis with hydroxychloroquine) and 2) participation in COVID-19 drug trials during ICU admission
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Any uncontrolled or significant concurrent illness that would put the patient at a greater risk or limit compliance with the study requirements

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Disease severity | on day 7
  Disease severity on the 7-point Ordinal World Health Organization (WHO) scale (for the current study, score 0 will be omitted and score 6 and 7 will be combined). The ordinal scale measures illness severity over time. This endpoint has been suggested by WHO for clinical trials in patients with COVID-19.

SECONDARY OUTCOMES:
Time to clinical improvement | within 14 days after enrolment
  Time to clinical improvement (time from randomisation to an improvement of two points on the seven-category WHO ordinal scale or live discharge from hospital, whichever came first)
Proportion of participants alive and not having required invasive or non-invasive ventilation | at 14 days after enrolment
  Proportion of participants alive and not having required invasive or non-invasive ventilation
Proportion of subjects with an ALI (defined by PaO2/FiO2 ratio of <300mmHg) | within 14 days after enrolment
  Proportion of subjects with an ALI (defined by PaO2/FiO2 ratio of <300mmHg)

OTHER OUTCOMES:
Changes in the ordinal WHO scale | from baseline over 14 days
  Changes in the ordinal WHO scale
Length of hospital stay in survivors | until day 28
  Length of hospital stay in survivors
Proportion of participants progressing to mechanical ventilation | on day 7 and day 14
  Proportion of participants progressing to mechanical ventilation
Proportion of participants requiring ICU treatment | on day 7 and 14
  Proportion of participants requiring ICU treatment
Length of ICU stay | until day 28
  Length of ICU stay
28 Ventilator-free days | until day 28
  28 Ventilator-free days
All-cause mortality | time from randomisation to death within four weeks
  All-cause mortality
Changes in biomarker level CRP (mg/l) | until day 14
  Changes in biomarker level CRP
Changes in biomarker level LDH (U/l) | until day 14
  Changes in biomarker level LDH
Changes in biomarker level D- Dimer (yg/ml) | until day 14
  Changes in biomarker level D-Dimer
Changes in biomarker level Ferritin (ng/ml) | until day 14
  Changes in biomarker level Ferritin
Changes in biomarker level Interleukin 6 (IL- 6) (pg/ml) | until day 14
  Changes in biomarker level IL-6
Changes in lymphocyte count (cells per microliter of blood) | until day 14
  Changes in lymphocyte count
Time to virological clearance of SARS-CoV-2 by PCR from upper or lower respiratory tract samples | time from enrolment to first of 2 negative assays at least 12 hours apart
  Time to virological clearance of SARS-CoV-2 by PCR from upper or lower respiratory tract samples
Proportion of patients receiving additional anti-inflammatory treatment such as tocilizumab or immunoglobulins | within 14 days
  Proportion of patients receiving additional anti-inflammatory treatment such as tocilizumab or immunoglobulins
Time to defervescence (temperature <38.0°C) | sustained for at least 48 hours
  Time to defervescence (temperature <38.0°C)
Time to clinical improvement (defervescence, normalization of oxygen saturation (>93%) and respiratory rate) until day 28 | until day 28
  Time to clinical improvement (defervescence, normalization of oxygen saturation (>93%) and respiratory rate)
Duration of supplemental oxygen | until day 28
  Duration of supplemental oxygen
Change in pharmacokinetics of conestat alfa | at baseline, day 1, day 3, day 7, day 10 (during admission) and day 14 (1/- 2days) or discharge date
  Peak serum concentration of conestat alfa will be measured
Change in pharmacodynamics of conestat alfa (C1-inhibitor (CI-INH) concentration) | at baseline, day 1, day 3, day 7, day 10 (during admission) and day 14 (1/- 2days) or discharge date
  Change in pharmacodynamics of conestat alfa (C1-inhibitor (CI-INH) concentration)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Osthoff, PD Dr. med., Principal Investigator — University Hospital Basel, Division of Internal Medicine
Locations (5):
- Práxis Pesquisa Medica, São Paulo, Brazil
- Hospital Universitario "Dr. José Eleiterio González", Colinia Mitras Centro, Monterrey, Nuevo Leon Mexico, Mexico
- Switzerland (3):
  - University Hospital Basel, Division of Internal Medicine, Basel
  - Kantonsspital St. Gallen, Klinik für Infektiologie/Spitalhygiene, Sankt Gallen
  - Stadtspital Triemli, Departement Innere Medizin, Zurich

REFERENCES:
- [Derived] Urwyler P, Leimbacher M, Charitos P, Moser S, Heijnen IAFM, Trendelenburg M, Thoma R, Sumer J, Camacho-Ortiz A, Bacci MR, Huber LC, Stussi-Helbling M, Albrich WC, Sendi P, Osthoff M. Recombinant C1 inhibitor in the prevention of severe COVID-19: a randomized, open-label, multi-center phase IIa trial. Front Immunol. 2023 Oct 27;14:1255292. doi: 10.3389/fimmu.2023.1255292. eCollection 2023. PMID 37965347
- [Derived] Urwyler P, Charitos P, Moser S, Heijnen IAFM, Trendelenburg M, Thoma R, Sumer J, Camacho-Ortiz A, Bacci MR, Huber LC, Stussi-Helbling M, Albrich WC, Sendi P, Osthoff M. Recombinant human C1 esterase inhibitor (conestat alfa) in the prevention of severe SARS-CoV-2 infection in hospitalized patients with COVID-19: A structured summary of a study protocol for a randomized, parallel-group, open-label, multi-center pilot trial (PROTECT-COVID-19). Trials. 2021 Jan 4;22(1):1. doi: 10.1186/s13063-020-04976-x. PMID 33397449